CLINICAL TRIAL: NCT04483856
Title: Efficacy and Tolerability Evaluation of a Topical Medical Device Based on SHBF in Management of Radiodermatitis. An Observer-masked, Controlled Study.
Brief Title: Efficacy and Tolerability Evaluation of a Topical MD Based on SHBF in Management of Radiodermatitis.
Acronym: DRESDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife Italia S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RELI/19/Der-Rdt/001
Record Dates: First submitted 2020-07-13; First posted 2020-07-23 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Radiodermatitis; Dermatitis, Radiation-Induced
Keywords: Radiodermatitis; DermoRelizema cream; DRESDA; Sodium Hyaluronate Butyrate Formiate; RELIFE
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Intervention Model Description: This is a post marketing, interventional, randomized, single-center, prospective, controlled study. Assessments and evaluations will be performed by a physician in a blind fashion.
Who Masked: Outcomes Assessor
Masking Description: Assessments and evaluations will be performed by a physician in a blind fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DermoRelizema cream (Experimental): The treatment will be applied since about 7 (±3) days prior to RT start and will continue until 14 days post RT end
  Interventions: Device: DermoRelizema cream
- Dexeryl (Active Comparator): The treatment will be applied since 7 (±3) days prior to RT start and will continue until 14 days post RT end (98-112 applications in total).
  Interventions: Device: Dexeryl

INTERVENTIONS:
Device: DermoRelizema cream — Fingertip units (FTU) depending from the extent of the affected skin to treat, two times per day for 7 (±3) days prior RT until about 14 (±3) days post RT end. The product can be used for further 2 weeks (from V3 to V4) in case of need, according to the investigator's judgment
  Arms: DermoRelizema cream
Device: Dexeryl — FTUs depending on the extent of the affected skin to treat, two times per day. The treatment will be applied since 7 (±3) days prior to RT start and will continue until 14 days post RT end (98-112 applications in total).
  Arms: Dexeryl

SUMMARY:
This is a post marketing, interventional, randomized, single-center, prospective, controlled study, for the evaluation of the clinical performance and tolerability of a cream-based medical device (DermoRelizemaTM cream) in the management care of radiodermatitis in women with breast cancer. Assessments and evaluations will be performed by a physician in a blind fashion.

The primary objective is Evaluation of the effects of DermoRelizemaTM cream in the management of the progression of RT-induced skin reactions and toxicity, using the grading system of the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/ EORTC), at the conclusion of the treatment period

DETAILED DESCRIPTION:
This is a post marketing, interventional, randomized, single-center, prospective, controlled study, for the evaluation of the clinical performance and tolerability of a cream-based medical device (DermoRelizemaTM cream) in the management care of radiodermatitis in women with breast cancer. Assessments and evaluations will be performed by a physician in a blind fashion.

The aim of this clinical study is to collect controlled evidences of the effectiveness and tolerability of DermoRelizemaTM cream in the management of RISRs in patients with breast cancer who will start the treatment with the product about one week before the start of RT.

The primary objective is Evaluation of the effects of DermoRelizemaTM cream in the management of the progression of RT-induced skin reactions and toxicity, using the grading system of the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/ EORTC), at the conclusion of the treatment period

ELIGIBILITY:
Inclusion Criteria:

* Women who give their written consent for participation in the study and willing to comply with all its procedures.
* Age ≥18 years.
* Women with breast cancer at any stage who have undergone quadrantectomy, for whom hypofractionated adjuvant RT of the thoracic region is indicated.
* RTOG/ EORTC radiodermatitis grade equal to 0 (zero) and good cutaneous trophism, in the region to be treated, according to investigator's judgement.
* Patients who are supposed to be cooperative with regard to compliance with study-related constraints.

Exclusion Criteria:

* Pregnant or lactating women (as not eligible to RT), and fertile women not following, at the investigators' judgement, an adequate contraceptive method.
* Subjects incapable of giving consent.
* Concomitant inflammatory skin diseases in acute phase such as: atopic dermatitis, contact dermatitis, psoriasis, lichen planus, pityriasis rosea.
* Collagen vascular disease, vasculitis, scleroderma, dermatomyositis, or systemic lupus erythematosus.
* Unhealed surgical sites, breast infections.
* Bilateral breast cancer or multiple neoplasia needing other independent RT treatments.
* Prior breast reconstructions, implants, and/or expanders.
* Known radio-sensitivity syndromes (e.g. ataxia-telangiectasia).
* Known history of intolerance or hypersensitivity to any ingredient of the study products.
* Previous RT in the same or different location.
* Topical pharmacological and medical device treatments on the skin region affected by the RT, in the last 2 weeks.
* Systemic or topical (including inhaled or intranasal) treatments containing corticosteroids of any class in the 2 days preceding the enrolment.
* Photo-therapy (PUVA, UVB) in the 2 weeks preceding the enrolment and/or planned to be administered during the course of the study.
* Participation in another clinical trial at the time of the randomization or within 28 days before randomization.
* Patient's difficulties or problems, in the judgment of the investigator, in being compliant with study procedures and requirements, including social or mental constrains.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patient with breast cancer
Enrollment: 70 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Francomano, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Modena University Hospital, Modena, Italy

IPD SHARING:
Plan to Share IPD: No
confidential information as per internal procedure of the Sponsor

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DermoRelizema Cream | Dexeryl
Started | 35 | 35
Completed | 31 | 30
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DermoRelizema Cream | Dexeryl | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.11 (10.86) | 59.56 (9.43) | 59.34 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 30 | 61
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression of Radio Therapy Induced Skin Reaction
Description: Evaluation of the effects of DermoRelizemaTM cream in the management of the progression of RT-induced skin reactions and toxicity
Time Frame: two weeks after the last RT sessiont,day 35-42
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 35 | 35
Participants | 35 | 33

2. Secondary Outcome: Progression of Radio Therapy-induced Skin Reactions Using the Grading System of the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Description: 1. Evaluation of the effects of DermoRelizemaTM cream, in the management of the progression of RT-induced skin reactions and toxicity, using the (RTOG/ EORTC) at the conclusion of the radiotherapy treatment (V2) and at study end (V4)
Time Frame: at the conclusion of the radiotherapy treatment, day 21-28 and at the study end day 49-56, reported day 56
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 30 | 31
Participants | 27 | 26

3. Secondary Outcome: Evaluation of the Radiation Symptoms (0 Best Result, 40 Worst Results)
Description: Evaluation of dermatitis symptoms management
Time Frame: up to 1 year
Population: Number of patients that are better on the radiation symptoms reported by the patient in a diary
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 30 | 31
units on a scale
  pain | 15.56 (15.58) | 17.90 (14.05)
  itch | 14.42 (10.29) | 15.79 (10.81)
  burning | 15.53 (11.97) | 12.65 (10.21)
  tenderness | 8 (9.28) | 12.96 (9.58)

4. Secondary Outcome: Severity of Radio Therapy-induced Skin Reactions Using the Grading System of the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Description: Evaluation of the severity of radiation dermatitis by the investigator using the RTOG/ EORTC (system of the Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer(grade 0-1: treatment is succesfull, grade 1 or magior: treatment insuccesful) ), at visits 2, 3 and 4
Time Frame: all study visits, day 21-28, day 35-42 and at the study end (day 49-56)
Population: Evaluation of the severity of radiation dermatitis by the investigator
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 31 | 28
Participants
  V2 no erythema | 9 | 2
  V2 erythema grade 1 | 18 | 24
  V2 erythema grade 2 | 4 | 1
  V2 erythema grade 3 | 0 | 1
  V3 no erythema | 16 | 9
  V3 erythema grade 1 | 13 | 18
  V3 erythema grade 3 | 1 | 1
  V4 no erythema | 29 | 25
  V4 erythema grade1 | 1 | 3

5. Secondary Outcome: Severity of Radiation Dermatitis With Radiation Dermatitis Severity (RDS) Scoring Scale
Description: Evaluation of the severity of radiation dermatitis by the investigator using the Radiation Dermatitis Severity (RDS) scoring scale. The severity of radiation dermatitis was measured using this scoring system, range 0.0 to 4.0 at increments of 0.5. The RDS score incorporates changes in redness, pigment, texture and integrity of the skin ( grade 0: best result, grade 4§: worst result)
Time Frame: all study visits, day 21-28, day 35-42 and at the study end (day 49-56)
Population: Evaluation of the severity of radiation dermatitis by the investigator
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 30 | 28
Participants
  V1 skin healthy | 30 | 28
  V4 grade 0 | 29 | 25

6. Secondary Outcome: Number of Participants With Progression of Radio Therapy Induced Skin Reaction
Description: Objective instrumental assessments of skin damage vascular parameters, tissue integrity and structural parameters,
Time Frame: all study visits, day 21-28, day 35-42 and at the study end (day 49-56)
Population: instrumental assessments of skin damage vascular parameters, tissue integrity and structural parameters
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 30 | 28
Participants | 30 | 28

7. Secondary Outcome: Patient Opinion on Cream With a Likert Scale
Description: Overall patient's opinion on the products' pleasantness
Time Frame: up to 1 year
Population: patient's opinion on the products' pleasantness
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 30 | 28
Participants
  smell pleasant/very pleasant | 18 | 15
  texture pleasant/very pleasant | 30 | 27
  spreadability pleasant/very pleasant | 30 | 28
  satisfaction pleasant/very pleasant | 29 | 27

8. Secondary Outcome: Adherence to Treatment of Patients
Description: Patient's adherence to treatment on a diary's scale ( 10 points, in whitc: 1 is the best, 100 is the worst)
Time Frame: up to 1 year
Population: Patient's adherence to treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 31 | 28
units on a scale | 96.50 (7.98) | 97.50 (8.82)

9. Secondary Outcome: Occurrence of Adverse Events
Description: Occurrence of Adverse Events
Time Frame: up to 1 year
Population: Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Cream | Dexeryl
Number analyzed (Participants) | 31 | 28
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: the adverse events are not related to the treatment performed.
Arm/Group | DermoRelizema Cream | Dexeryl
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT04483856/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT04483856/SAP_001.pdf